CLINICAL TRIAL: NCT05335122
Title: A Prospective, Multi-center, Randomized, Parallel-group, Controlled Study to Evaluate the Efficacy and Safety of OTX-TIC (Travoprost) Intracameral Implant in Subjects With Open-angle Glaucoma (OAG) or Ocular Hypertension (OHT)
Brief Title: A Study to Evaluate the Efficacy and Safety of OTX-TIC (Travoprost) Intracameral Implant for Patients With Open-angle Glaucoma (OAG) or Ocular Hypertension (OHT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OTX-TIC-2020-201
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Intervention Model Description: Parallel: Participants are assigned to one of three groups in parallel for the duration of the study
Who Masked: Participant, Outcomes Assessor
Masking Description: Sponsor, Study Coordinator, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OTX-TIC Low Dose (Experimental): Travoprost Intracameral Implant low dose
  Interventions: Drug: OTX-TIC low dose Travoprost Intracameral Implant
- OTX-TIC High Dose (Experimental): Travoprost Intracameral Implant high dose
  Interventions: Drug: OTX-TIC high dose Travoprost Intracameral Implant
- Durysta (Active Comparator): Bimatoprost Intracameral Implant 10 µg
  Interventions: Drug: Durysta, Bimatoprost Intracameral Implant 10 µg

INTERVENTIONS:
Drug: OTX-TIC low dose Travoprost Intracameral Implant — OTX-TIC implant is injected into the anterior chamber of the eye.
  Arms: OTX-TIC Low Dose
Drug: OTX-TIC high dose Travoprost Intracameral Implant — OTX-TIC implant is injected into the anterior chamber of the eye.
  Arms: OTX-TIC High Dose
Drug: Durysta, Bimatoprost Intracameral Implant 10 µg — Durysta is injected into the anterior chamber of the eye.
  Arms: Durysta

SUMMARY:
To assess efficacy, and safety of a single sustained release dose of the OTX-TIC drug product (2 travoprost dose strengths) in subjects with Open Angle Glaucoma (OAG) or Ocular Hypertension (OHT)

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, parallel-group, controlled study to evaluate the efficacy, and safety of OTX-TIC (travoprost) intracameral implant in subjects with open angle glaucoma (OAG) or ocular hypertension (OHT). Approximately 105 subjects will be enrolled in this study at approximately 20 sites in the US. Subjects will be a randomized to one of three treatment groups OTX-TIC drug product (2 travoprost dose strengths) compared to a single injection of DurystaTM. Non study eyes will be treated with the PGA, if not contraindicated.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years of age or older at the time of screening
* Provide written informed consent and are able to comply with all study requirements
* Are willing to withhold glaucoma medications according to the study requirements, and in the opinion of the investigator can do so without significant risk
* Have a negative pregnancy test result for women of childbearing potential at Baseline
* Have a documented diagnosis of OHT, or OAG in the study eye

Exclusion Criteria:

* Have an uncontrolled systemic disease or a debilitating disease (e.g., cardiovascular, hypertension, uncontrolled diabetes)
* Are currently pregnant or breast-feeding or of childbearing potential without the use of adequate contraceptive methods during the length of the study
* Non-responsive to topical prostaglandins, prostamides or prostaglandin analogs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Efficacy Outcome: IOP changes from Baseline | Diurnal IOP [Time Frame: diurnal IOP at the 2 Week Visit] Diurnal IOP [Time Frame: diurnal IOP at the 6 Week Visit] Diurnal IOP [Time Frame: diurnal IOP at the 12 Week Visit]
  IOP changes from baseline at 8AM, 10AM, and 4PM at Week 2, Week 6, and Week 12 in the study eye

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Ocular Therapeutix, Inc., Dothan, Alabama
  - Ocular Therapeutix, Inc., Huntington Beach, California
  - Ocular Therapeutix, Inc., Irvine, California
  - Ocular Therapeutix, Inc., Los Angeles, California
  - Ocular Therapeutix, Inc., Pasadena, California
  - Ocular Therapeutix, Inc., Petaluma, California
  - Ocular Therapeutix, Inc., Redlands, California
  - Ocular Therapeutix, Inc., Torrance, California
  - Ocular Therapeutix, Inc., Clearwater, Florida
  - Ocular Therapeutiux, Inc., Delray Beach, Florida
  - Ocular Therapeutix, Inc., Fort Myers, Florida
  - Ocular Therapeutix, Inc., Roswell, Georgia
  - Ocular Therapeutix, Inc., Rock Island, Illinois
  - Ocular Therapeutix Inc, Carmel, Indiana
  - Ocular Therapeutix, Inc., Saint Joseph, Michigan
  - Ocular Therapeutix, Inc., Saint Joseph, Missouri
  - Ocular Therapeutix Inc., St Louis, Missouri
  - Ocular Therapeutix, Inc., Dover, New Jersey
  - Ocular Therapeutix, Inc., Troy, New York
  - Ocular Therapeutix, Inc., Durham, North Carolina
  - Ocular Therapeutiux, Inc., Fargo, North Dakota
  - Ocular Therapeutix, Inc., Cleveland, Ohio
  - Ocular Therapeutix Inc, Oklahoma City, Oklahoma
  - Ocular Therapeutix, Inc., Cranberry Township, Pennsylvania
  - Ocular Therapeutix, Inc., Philadelphia, Pennsylvania
  - Ocular Therapeutix, Inc., Austin, Texas
  - Ocular Therapeutix, Inc., Dallas, Texas
  - Ocular Therapeutix, Inc., El Paso, Texas
  - Ocular Therapeutix, Inc., Houston, Texas
  - Ocular Therapeutix, Inc., Kenosha, Wisconsin